CLINICAL TRIAL: NCT00000206
Title: Clinical Rescue Protocol
Brief Title: Clinical Rescue Protocol - 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-06082-2; R18DA006082 (NIH); R18-06082-2
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-11

CONDITIONS: Opioid-Related Disorders
Keywords: Opioid
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine

SUMMARY:
The purpose of this study is to detect increasing medication dose results in heroin cessation for patients still using, to determine if decreasing medication dose in patients unable to tolerate medication dose increases retention, and to determine if blood levels of methadone or buprenorphine correlate with clinical response.

ELIGIBILITY:
Inclusion Criteria:

M/F ages 21-50. Opiate dependence according to DSM-IV criteria. Self-reported use within the last 30 days. Agreeable to conditions of study and signed informed consent.

Exclusion Criteria:

Psychiatric disorder that requires medication therapy. History of seizures. Pregnant and/or nursing women. Dependence on ETOH or benzodiazepines or other sedative-hynotics. Acute hepatitis. Other medical conditions that deem participation to be unsafe.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1991-04; Primary Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Retention
Opiate use
Opiate craving
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Walter Ling, M.D., Principal Investigator — Friends Research Institute, Inc.
Locations (1):
- Friends Research Institute, Los Angeles, California, United States

REFERENCES:
- [Background] Ling W, Shoptaw S, Wesson D, Rawson RA, Compton M, Klett CJ. Treatment effectiveness score as an outcome measure in clinical trials. NIDA Res Monogr. 1997;175:208-20. No abstract available. PMID 9467800